CLINICAL TRIAL: NCT05300750
Title: The Effect of Post Cesarean Section Protocol of Care on Early and Follow up Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rania Mahmoud Abdel Ghani, Assisstant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: No.15-2019
Record Dates: First submitted 2022-03-02; First posted 2022-03-29 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Cesarean Section
Keywords: Oral fluid; Chewing gum; Post cesarean; Intestinal movement; Passage of flatus
MeSH Terms: interventions — Fluid Therapy; Chewing Gum

STUDY DESIGN:
Intervention Model Description: Randomized controlled trail (Parallel group design) is an experimental study design in which each subject is randomized to one of two or more distinct treatment/intervention groups. Those who are assigned to the same treatment are referred to as a treatment group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral Fluid (Experimental): The oral fluid intake was in form of peppermint or anise
  Interventions: Other: Oral fluids
- Chewing Gum (Experimental): Free sugar gum
  Interventions: Other: Chewing gum
- Standard hospital care (No Intervention): Control group

INTERVENTIONS:
Other: Oral fluids — Starting amount of oral fluid after 2 hours post C/s should be 5cm and then increase gradually to be 45-50 cm of oral fluid at 4 hours post C/s and 100 cm each hours later.
  Arms: Oral Fluid
Other: Chewing gum — Chewed free sugar gum for 15 minutes
  Arms: Chewing Gum

SUMMARY:
The aim of the current study is to evaluate the effect of post cesarean section protocol of care on early and follow up outcomes.The criteria for inclusion were; mothers can read and write, primipara or multipara who was admitted to postpartum unit, age ranged between 20-35 years, under epidural anesthesia, gestational age (≥ 37 weeks) newborn, uncomplicated elective or under C/s for abnormal lie, abnormal presentation, cephalo- pelvic disproportion. Mothers with any medical disorders or post C/s complications were excluded from the present study.Two post C/s regimens were approached for two groups of interventions; 1) oral fluids group (A) and 2) chewing gum group (B) versus standard hospital care group (C). Both interventions groups (A&B) received early ambulation, breathing and coughing exercises protocol of care besides. Both groups of intervention received the proposed protocol at 2, 4, 6 hours post -cesarean.

Regarding to the intervention group (A) in which mothers received oral fluid, the starting amount of fluid after 2 hours post C/s should be 5cm and then increase gradually to be 45-50 cm of oral fluid at 4 hours post C/s and 100 cm each hours later. The oral fluid intake was in form of peppermint or anise. While in the intervention group (B), mothers chewed free sugar gum for 15 minutes in the same time points of group (A) at 2, 4 and 6 hours after C/s. Further, ambulation of mothers started after four hours post C/s.

Furthermore, before discharge both intervention groups were received booklet contained health education for healthy diet with balanced meal, different position for breast feeding, dealing with C/s wound, dealing with post C/s minor discomfort, information related to postpartum danger signs (i.e. foul vaginal discharge, sever incision pain, discharge from suture line, painful calf muscle, burning sensation on urination, heavy vaginal bleeding, symptoms of anxiety. Further, each mother had been informed that if any minor discomforts or any danger signs appeared and couldn't deal with, contact the researcher directly to help in management and referral with available phone numbers. Also, each mother was informed to come for obligatory postpartum clinic for follow up on day 10 after cesarean section for complete check and follow up.

DETAILED DESCRIPTION:
The aim of the current study is to evaluate the effect of post cesarean section protocol of care on early and follow up outcomes. The criteria for inclusion were; mothers can read and write primipara or multipara who was admitted to postpartum unit, age ranged between 20-35 years, under epidural anesthesia, gestational age (≥ 37 weeks) newborn, and uncomplicated elective or under C/s for abnormal lie, abnormal presentation, cephalo- pelvic disproportion. Mothers with any medical disorders or post C/s complications were excluded from the present study. An ethical approval was obtained from the ethical research committee of the faculty of nursing, (No.15-2019). As well as, an official permission was taken from authoritative personnel at obstetrics and gynecology hospital and postpartum department to conduct the study The researcher introduced herself to the post C/s mothers who met the inclusion criteria and informed them about the purpose and nature of the study to obtain their acceptance to participate in the study, all the mothers were informed that participation in the study is voluntary and they could withdraw from the study at any time without any negative consequences. Written consent was obtained prior to the commencement of data collection. Anonymity and confidentiality related to the information to the identity of each post C/s mothers were kept in a locked file. File folder was identified only by numbers; also, recorded data were assured through coding of data and assuring that. An official permission for conducting this study was obtained from the administrative authorities of El Kasr El Aini hospitals. Gathering data took place from the period of May 2019 up to November 2020. Six cases/weak for 25 weeks (i.e. the Covid -19 condition disturbed the continuity of the process). Recruitment of participant and Randomization Upon full evaluation and matching the diagnosis, all mothers who met the inclusion criteria were enrolled in the trial .randomization was achieved using randomly permuted blocks of different sizes (3, 6, and 9) .each block used for one time except block nine which repeated twice. The ratio of intervention groups versus the standard hospital care was 1:1:1 when the intervention group of oral fluid took symbol (A) and the intervention group of chewing gum took symbol (B) and the standard hospital care group took symbol (C) for the distribution of permuted blocks .the permuted blocks 3disturbuted 18 cases, .the permuted blocks 6 distributed 36cases, while the permuted blocks 9 distributed 54 cases and repeated twice up till the total number of sample was reached (I.e. 150). Concealed opaque envelopes with sequential numbers were utilized. A team of two clinical instructors who were trained in the maternal and newborn health nursing department were shared in the allocation of the mothers to different groups after receiving the appropriate training. Mothers, who met the inclusion criteria, were assigned to the interventions groups or the control group .utilizing the sequential opaque envelops. The main researcher was outside the process of allocation. Blinding and masking: Regarding the nature of the intervention there were difficulties in masking both the participant and the researcher. The researcher interviewed the mothers, explained the purpose of the study and written consent was obtained. Mothers were assured that their participation in the study was voluntary and that privacy and confidentiality were ensured. Baseline data of demographic characteristic and obstetrical history were gathered. In addition to the intestinal movement sound, passing of flatus, presence of nausea or vomiting .which carried two hours after cesarean section. Two post C/s regimens were approached for two groups of interventions; 1) oral fluids group (A) and 2) chewing gum group (B) versus standard hospital care group (C). Both interventions groups (A&B) received early ambulation, breathing and coughing exercises protocol of care besides. Both groups of intervention received the proposed protocol at 2, 4, 6 hours post -cesarean. Regarding to the intervention group (A) in which mothers received oral fluid. The starting amount of fluid after 2 hours post C/s should be 5cm and then increase gradually to be 45-50 cm of oral fluid at 4 hours post C/s and 100 cm each hours later. The oral fluid intake was in form of peppermint or anise. While in the intervention group (B), mothers chewed free sugar gum for 15 minutes in the same time points of group (A) at 2, 4 and 6 hours after C/s. Further, ambulation of mothers started after four hours post C/s.

Furthermore, before discharge both intervention groups were received booklet contained health education for healthy diet with balanced meal, different position for breast feeding, dealing with C/s wound, dealing with post C/s minor discomfort, information related to postpartum danger signs (i.e. foul vaginal discharge, sever incision pain, discharge from suture line, painful calf muscle, burning sensation on urination, heavy vaginal bleeding, symptoms of anxiety. Further, each mother had been informed that if any minor discomforts or any danger signs appeared and couldn't deal with, contact the researcher directly to help in management and referral with available phone numbers. Also, each mother was informed to come for obligatory postpartum clinic for follow up on day 10 after cesarean section for complete check and follow up. Two stages of follow up; first: evaluation of the intervention's effect at hospital and before discharge. Second: follow up of mothers at home. First: evaluation of the intervention effect: In this stage as described before all mothers in both intervention groups received the planned protocol of care (i.e. oral fluids or gum besides the ambulation and breathing exercises), and had been evaluated for intestinal sound, passage of flatus, and timing of breast feeding at the time points of 4, 6 and 8 hours post cesarean section. Second: follow up of mothers at home: In this stage, mothers were followed at third, seventh days post-cesarean section at home by phone. The researcher assessed their abilities to carry their routine and daily activities as well as ensured that there were no complication appeared or re-hospitalization occurred. Further at ten days post cesarean section, each mother came to postpartum clinic in order to check the wound condition and overall health condition and removed the C.S. sutures.

ELIGIBILITY:
Inclusion Criteria:

Mothers can read and write

* Primipara or multipara who was admitted to postpartum unit
* Age ranged between 20-35 years
* Under epidural anesthesia, gestational age (≥ 37 weeks) newborn
* Uncomplicated elective or under C/s for abnormal lie
* Abnormal presentation, cephalo- pelvic disproportion.

Exclusion Criteria:

- Mothers with any medical disorders or post C/s complications

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Mothers in postaprtum period
Enrollment: 150 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-02-27 (Actual)

PRIMARY OUTCOMES:
Intestinal sound | From 4hours post-cesarean section up to 8 hours later
  Hearing of intestinal sound after cesarean section after receiving the intervention (oral fluid or chewing gum, two hours post ceserean section).
  Measured by post cesarean section early assessment sheet. This tool divided into three parts; part (1) includes base line data of the mothers such as physiological condition after 2 hours post Cs delivery (vital signs, intestinal movement, passage the flatus, abdominal distension, nausea, vomiting, and colic related to distention). Part: (2) includes data related to assessment of mothers condition after first ambulation 4 hours post Cs delivery (i.e. the time of early ambulation, feeling of drowsiness in change position from sitting to standing or walking, ability to walk, ability to sit;. While the third part includes assessment of mothers' abilities to do breathing exercises.
Passage of flatus | From 4hours post-cesarean section up to 8 hours later
  Assessment of passage of flatus after receiving the intervention (oral fluid or chewing gum, two hours post ceserean section).
  Measured by post cesarean section early assessment sheet. This tool divided into three parts; part (1) includes base line data of the mothers such as physiological condition after 2 hours post Cs delivery (vital signs, intestinal movement, passage the flatus, abdominal distension, nausea, vomiting, and colic related to distention). Part: (2) includes data related to assessment of mothers condition after first ambulation 4 hours post Cs delivery (i.e. the time of early ambulation, feeling of drowsiness in change position from sitting to standing or walking, ability to walk, ability to sit;. While the third part includes assessment of mothers' abilities to do breathing exercises.
Duration of hospital stay | From 1 hour post-cesarean section up to 12 hours later
  Duration of hospital stay after cesarean section. It measured by numbers of hours started immediately after C/S operation up till the time of hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Shadia A Abdel Kader Hassan, Professor, Study Chair — Faculty of Nursing- Cairo University; Magda A Ahmed Fawaz, Professor, Study Director — Faculty of Nursing- Cairo University; Ahmed A Mahmoud Sayed, Professor, Study Director — Cairo University
Locations (1):
- Eman Said Abo El Ella Hassan, Faisal, Giza Governorate, Egypt